CLINICAL TRIAL: NCT04539899
Title: Evaluation of the Influence of the Virtual Reality Helmet on Pain During IUD Insertion : REAVIST
Brief Title: Evaluation of the Influence of the Virtual Reality Helmet on Pain During IUD Insertion
Acronym: REAVIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC20_8886_REAVIST
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: IUD

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR+ (Experimental): For patients in the experimental group, using the virtual reality helmet, the caregiver will position the helmet on the patient when she is placed on the gynecological examination table. He or she will make sure that the patient can see and hear the current sequence. The caregiver can then proceed with the different steps of the IUD insertion. Once the procedure is completed, the caregiver will indicate to the patient that she can remove the headphones.
  Interventions: Other: VR+
- VR- (No Intervention): For patients in the control group, without a helmet, the course of the consultation will not be modified.

INTERVENTIONS:
Other: VR+ — Use of a virtual reality helmet during IUD insertion
  Arms: VR+

SUMMARY:
Given the current lack of satisfactory options for the management of IUD insertion pain, could the virtual reality headset be an innovative and effective tool? The objective is to compare the pain experienced during IUD insertion between a group of women wearing a virtual reality helmet and a group not wearing one.

Observational, prospective, randomized, open-label, monocentric study.

ELIGIBILITY:
Inclusion Criteria:

* Female adult
* Who has benefited from contraceptive counseling
* The choice of an IUD (hormonal or copper)
* Having signed a written informed consent.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Pre-existing dizzying sensations
* Severe facial wounds
* History of epilepsy
* Persons of full age subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Method of female contraception
Enrollment: 100 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
NRS during IUD insertion | 20 minutes
  The assessment criterion used is the written self-report numerical scale (NRS) from 0 to 10 (0 = no pain, 10 = extremely painful)

SECONDARY OUTCOMES:
Stress level difference with virtual reality | 20 minutes
  Difference of stress between experimental and control group using self-assessment anxiety scale specially designed for the study, where 0 = non stress and 10 = maximum of stress
Satisfaction level difference with virtual reality | 20 minutes
  Difference of satisfaction between experimental and control group using self-assessment anxiety scale specially designed for the study, where 0 = not satisfied at all and 10 = totally satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France